CLINICAL TRIAL: NCT02650830
Title: Seum Bile Acid Profile in Type 2 Diabetes and Association Between Bile Cid Profile and Adipokine or Oxidative Stress
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2015-0503
Record Dates: First submitted 2016-01-06; First posted 2016-01-08 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Type 2 Diabetes; Prediabetes; Non-alcoholic Fatty Liver Disease; Metabolic Syndrome
Keywords: type 2 diabetes; prediabetes; bile acids profile; GLP-1; FGF-19
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Non-alcoholic Fatty Liver Disease; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum (blood), whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1) Normal control: metabolically healthy with no obesity
- 2) prediabetes: defined in 'inclusion criteria'
- 3) type 2 diabetes: defined in 'inclusion criteria'

SUMMARY:
"The goal of this work is to critically test the hypothesis that there exists a different profile of bile acids (BAs) in patient with type 2 diabetes mellitus (T2DM) compared with normal controls. Through confirmation of different profile of BAs in T2DM, investigator will suggest modulation of specific bile acids as a new possible treatment target in patients with T2DM. Investigator also expect the specific BAs signature will be used to screen T2DM before hyperglycemia.

In addition, investigator will evaluate the association between each BA species and serum total glucagon like peptide-1 (GLP-1) or fibroblast growth factor-19 (FGF-19) concentrations to determine if the specific BAs profile is related with total GLP-1 or FGF-19 concentration in serum. Investigatr also evaluates the correlation between each BA species and metabolic profiles and oxidative stress marker to find possible roles of each BA component in glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

1. pre-diabetes 1. defined according to the ADA guideline (prediabetes definition) FPG 100 mg/dL (5.6 mmol/L) to 125 mg/dL (6.9 mmol/L) (IFG) or 2-h PG in the 75-g OGTT 140 mg/dL (7.8 mmol/L) to 199 mg/dL (11.0 mmol/L) (IGT) or A1C 5.7-6.4% (39-46 mmol/mol)
2. type 2 diabetes 1. defined according to the ADA guideline (DM definition) FPG ≥126 mg/dL (7.0 mmol/L) or 2-h PG ≥200 mg/dL (11.1 mmol/L) in the 75-g OGTT or A1C ≥6.5% (48 mmol/mol) or In a patient with classic symptoms of hyperglycemia or hyperglycemic crisis, a random plasma glucose ≥200 mg/dL (11.1 mmol/L) or 2. taking any anti-diabetic medications
3. Normal control 1. should not be included in other groups as above and 2. not taking any medication related to diabetes and dyslipidemia and 3. BMI <25kg/m2

Exclusion Criteria:

1. subjects who refused to agree with informed consents
2. subjects with organ-transplantation
3. pregnant women
4. type 1 diabetes -

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects are recruited from either patients who visit out-patient clinics (Diabetes center in Severance hospital) or healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2015-09-12 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
bile acid profile | 8h fasting blood sample
  Bile acids profile to predict T2DM will be measured using high performance liquid chromatography-tandem mass spectrometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
no plan to share data